CLINICAL TRIAL: NCT05483075
Title: An Exploratory Study Evaluating the Feasibility of a Health Care Provider Guided Exercise Intervention Prior to Surgical Resection of Pancreatic Cancer With Biological Correlative Studies
Brief Title: Feasibility of a Health Care Provider Guided Exercise Intervention Prior to Surgical Resection of Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-00289
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer
Keywords: HCP-Guided Exercise
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCP-Guided Exercise (Experimental): Participants will schedule twice-weekly in-person visits to conduct health care provider (HCP)-supervised exercise activity for a minimum of 30 minutes. At least 3 additional times per week, participants will conduct self-directed exercise at home. Activity and other outcomes will be monitored with an Actigraph Centrepoint Insight Watch.
  The HCP guided therapy will continue on a weekly basis for at least 2 weeks and up to a maximum of 4 weeks.
  Interventions: Behavioral: HCP-Guided Exercise Training Program
- Control (No Intervention): Participants will not participate in the HCP-guided exercise intervention but will wear the Actigraph Centrepoint Insight Watch.

INTERVENTIONS:
Behavioral: HCP-Guided Exercise Training Program — Individually tailored exercise program consisting of aerobic training (5 days per week for a minimum of 30 minutes at moderate intensity) and strength training (2 days per week at moderate intensity).
  Two days per week the participant will receive their exercise program at NYU Langone Health. When at NYU, the training will be supervised by a physical therapist and will consist of the following: warm-up of 5 minutes, 30 minutes of aerobic exercise on either a stationary bike or treadmill at 60-70% of maximum heart rate. Following aerobic training, strength training will be carried out. Strength training will consist of 1 exercise per major muscle group, 8-12 reps, 1-3 sets at moderate intensity.
  The remaining three days a week the participant will perform aerobic training at home by exercising on a bicycle or by walking fast for a minimum of 30 mins at moderate intensity (60-70% of max HR).
  Arms: HCP-Guided Exercise

SUMMARY:
Pilot study evaluating the feasibility of a 2-4 week health care provider guided exercise intervention prior to surgery for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to participate in the study procedures
2. Pathologically confirmed pancreatic cancer
3. Candidate for neoadjuvant therapy followed by surgical resection with potentially curative intent. Note: There is no limitation on duration of neoadjuvant therapy.
4. Planned to have at least 2 weeks after completing the last neoadjuvant therapy and surgery
5. Over the age of 18
6. Ability to engage in physical activity as determined by physiatrist review after completion of the Physical Activity Readiness questionnaire (PAR-Q) exercise survey and chart review
7. Agree to study blood draws and tissue collection

Exclusion Criteria:

1. Evidence of metastatic disease
2. Inability to complete physical activity due to recent injury or surgery
3. Uncontrolled heart disease limiting physical activity
4. Participation in another interventional trial that excludes participation in this protocol
5. Subjects who anticipate undergoing a procedure during the course of the trial that will render them unable to engage in physical activity for more than 48 hours
6. Pregnant subjects
7. Individuals who lack the capacity to consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Number of Intervention Arm Participants in Compliance with HCP Exercise Intervention | Up to Week 4
  Compliance with HCP exercise intervention is defined as successful completion of at least 150 minutes of weekly moderate-to-intense physical activity over a minimum of 2 weeks for every week of the prescribed intervention (2, 3 or 4 weeks).

SECONDARY OUTCOMES:
Number of Participants who Experience Adverse Events (AEs) | Up to Week 4
  AEs defined as any symptom, sign, illness or experience that develops or worsens in severity during the course of the study.
Number of Participants who Experience an Event that Leads to Delay in Surgical Resection | Up to Week 4
Change in Number of Tumor-Infiltrating CD8-Positive T Cells | Baseline, Final Study Visit (Between Weeks 2-4)
  Multiplex immune-fluorescence staining conducted on tumor tissue samples to assess number of cluster designation 8 (CD8)-positive T cells.
Change in Number of Tumor-Infiltrating CD8-Positive T Cells Expressing IL-15Ra | Baseline, Final Study Visit (Between Weeks 2-4)
  Multiplex immune-fluorescence staining conducted on tumor tissue samples to assess number of CD8-positive T cells expressing Interleukin 15 Receptor Alpha Subunit (IL-15Ra).
Change in Number of Tumor-Infiltrating CD8-Positive T Cells Expressing GZMB | Baseline, Final Study Visit (Between Weeks 2-4)
  Multiplex immune-fluorescence staining conducted on tumor tissue samples to assess number of CD8-positive T cells expressing Granzyme B (GZMB).
Change in Number of Tumor-Infiltrating CD8-Positive T Cells Expressing CD3 | Baseline, Final Study Visit (Between Weeks 2-4)
  Multiplex immune-fluorescence staining conducted on tumor tissue samples to assess number of CD8-positive T cells expressing cluster designation 3 (CD3).
Change in Number of Circulating CD8-Positive T Cells Expressing IL-15Ra as Assessed by Flow Cytometry | Baseline, Final Study Visit (Between Weeks 2-4)
  Flow cytometry conducted on patient blood samples to assess number of circulating CD8-positive T cells expressing Interleukin 15 Receptor Alpha Subunit (IL-15Ra).
Time Spent in Moderate-to-Vigorous Physical Activity (MVPA) | Up to Week 4
  Monitored using the ActiGraph Centrepoint Insight Watch in conjunction with ActiLife software and validated algorithms.
  Moderate Activity is defined as between 3.00 and 5.99 metabolic equivalents (METs). Vigorous Activity is defined as at least 6.00 METs. MET is defined as the ratio of the work metabolic rate to the resting metabolic rate.
Time Spent in Sedentary Behavior | Up to Week 4
  Monitored using the ActiGraph Centrepoint Insight Watch in conjunction with ActiLife software and validated algorithms.
  Sedentary Behavior is defined as less than 0.11 metabolic equivalents (METs). MET is defined as the ratio of the work metabolic rate to the resting metabolic rate.
Average Daily MET Rates | Up to Week 4
  Monitored using the ActiGraph Centrepoint Insight Watch in conjunction with ActiLife software and validated algorithms.
  MET is defined as the ratio of the work metabolic rate to the resting metabolic rate. Light intensity activities are defined as less than 3 METs, moderate intensity activities are defined as between 3 and 5.99 METs, and vigorous intensity activities are defined as 6 METs or greater.
Total Physical Activity Energy Expenditure | Up to Week 4
  Monitored using the ActiGraph Centrepoint Insight Watch in conjunction with ActiLife software and validated algorithms. Expressed in kcal/day.
Minutes Spent in Rapid Eye Movement (REM) Sleep | Up to Week 4
  Monitored using ActiGraph Centrepoint Insight Watch.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Oberstein, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Health Ambulatory Care Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to:
  Paul Oberstein 212-731-6120 paul.oberstein@nyulangone.org
  The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to paul.oberstein@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.